CLINICAL TRIAL: NCT00038467
Title: Randomized Double-Blind Trial In Postmenopausal Women With Primary Breast Cancer Who Have Received Adjuvant Tamoxifen For 2-3 Years, Comparing Subsequent Adjuvant Exemestane Treatment With Further Tamoxifen
Brief Title: Randomized Trial Of Exemestane Versus Continued Tamoxifen In Postmenopausal Women With Early Breast Cancer
Acronym: IES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: International Collaborative Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96-OEXE-031; A5991012
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; exemestane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator)
  Interventions: Drug: Tamoxifen
- A (Experimental)
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen 20 mg/day tablets administered p.o. for a period ranging from 2.5 to 3 years.
  Arms: B
Drug: Exemestane — Exemestane 25 mg/day tablets administered p.o. for a period ranging from 2.5 to 3 years.
  Arms: A

SUMMARY:
To compare the sequential administration of exemestane with administration of further tamoxifen until 5 years in postmenopausal women with operable breast cancer who have already received 2-3 years of adjuvant tamoxifen, in terms of disease-free survival (DFS), overall survival (OS), incidence of contralateral breast cancer and long-term tolerability.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with histologically or cytologically confirmed primary breast adenocarcinoma, receiving tamoxifen and have been treated with tamoxifen continuously for between 2 and 3 years and one month, and still free of disease

Exclusion Criteria:

* unresectable breast cancer
* ER negative primary tumor

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4740 (Actual)
Dates: Start 1998-02; Primary Completion 2003-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (321):
- United States (39):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Green Valley, Arizona
  - Pfizer Investigational Site, Green Velley, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Fort Collins, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Thornton, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jacksonville Beach, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orange Park, Florida
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Latham, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Garland, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, McAllen, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Odessa, Texas
  - Pfizer Investigational Site, Pasadena, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Sherman, Texas
  - Pfizer Investigational Site, Sugar Land, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Weslaco, Texas
  - Pfizer Investigational Site, Spokane, Washington
- Argentina (8):
  - Pfizer Investigational Site, Haedo, Buenos Aires
  - Pfizer Investigational Site, San Isidro, Buenos Aires
  - Pfizer Investigational Site, San Martín, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
  - Pfizer Investigational Site, Rosario, Pcia. de Santa Fe
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Córdoba
- Australia (8):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Dubbo, New South Wales
  - Pfizer Investigational Site, Liverpool, New South Wales
  - Pfizer Investigational Site, Waratah, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Bendigo, Victoria
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Ringwood East, Victoria
- Belgium (18):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Arlon
  - Pfizer Investigational Site, Baudour
  - Pfizer Investigational Site, Brasschaat
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Haine-Saint-Paul
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Kraainem
  - Pfizer Investigational Site, La Louvière
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Merksem
  - Pfizer Investigational Site, Namur
  - Pfizer Investigational Site, Verviers
  - Pfizer Investigational Site, Wilrijk
- Pfizer Investigational Site, Sarajevo, Bosnia and Herzegovina
- Bulgaria (3):
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
- Croatia (3):
  - Pfizer Investigational Site, Osijek
  - Pfizer Investigational Site, Split
  - Pfizer Investigational Site, Zagreb
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Prague
- Denmark (10):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Esbjerg
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Herning
  - Pfizer Investigational Site, Hilleroed
  - Pfizer Investigational Site, Koebenhavn OE
  - Pfizer Investigational Site, Næstved
  - Pfizer Investigational Site, Roskilde
  - Pfizer Investigational Site, Vejle
  - Pfizer Investigational Site, Viborg
- Pfizer Investigational Site, Cairo, Egypt
- Pfizer Investigational Site, Tartu, Estonia
- France (26):
  - Pfizer Investigational Site, Bordeaux, France
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Annecy
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Évreux
  - Pfizer Investigational Site, Lagny-sur-Marne
  - Pfizer Investigational Site, Le Havre
  - Pfizer Investigational Site, Le Mans
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Meaux
  - Pfizer Investigational Site, Montbéliard
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Perpignan
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Cloud
  - Pfizer Investigational Site, Saint-Herblain
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
- Germany (17):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Gera
  - Pfizer Investigational Site, Greiz
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hildburghausen
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Riesa
  - Pfizer Investigational Site, Rodewisch
  - Pfizer Investigational Site, Saarbrücken
  - Pfizer Investigational Site, Suhl
  - Pfizer Investigational Site, Weiden
- Greece (2):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Heraklion, Crete
- Pfizer Investigational Site, New Territories, Hong Kong
- Pfizer Investigational Site, Budapest, Hungary
- Ireland (4):
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Cork, Ireland
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Galway
- Israel (5):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Kfar Saba
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Rehovot
- Italy (37):
  - Pfizer Investigational Site, Carpi, Modena
  - Pfizer Investigational Site, Alba (CN)
  - Pfizer Investigational Site, Aviano (PN)
  - Pfizer Investigational Site, Bergamo
  - Pfizer Investigational Site, Biella
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Casale Monferrato, AL
  - Pfizer Investigational Site, Correggio
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Cuneo
  - Pfizer Investigational Site, Fermo FM
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Lecco
  - Pfizer Investigational Site, Lodi
  - Pfizer Investigational Site, Mantova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Monserrato (CA)
  - Pfizer Investigational Site, Monza
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Piacenza
  - Pfizer Investigational Site, Pietra Ligure (SV)
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Reggio Emilia
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Terni
  - Pfizer Investigational Site, Thiene (VI)
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Tortona
  - Pfizer Investigational Site, Trescore Balneario BG
  - Pfizer Investigational Site, Treviglio (BG)
  - Pfizer Investigational Site, Varese
- Pfizer Investigational Site, Luxembourg, Luxembourg
- Pfizer Investigational Site, Floriana, Malta
- Netherlands (20):
  - Pfizer Investigational Site, Amersfoort
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Apeldoorn
  - Pfizer Investigational Site, Blaricum
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Delft
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Enschede
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Hengelo
  - Pfizer Investigational Site, Leeuwarden
  - Pfizer Investigational Site, Leiden
  - Pfizer Investigational Site, Leidschendam
  - Pfizer Investigational Site, Podybus 90153
  - Pfizer Investigational Site, Roermond
  - Pfizer Investigational Site, Sittard
  - Pfizer Investigational Site, The Hague
  - Pfizer Investigational Site, Utrecht
  - Pfizer Investigational Site, Veldhoven
  - Pfizer Investigational Site, Zaandam
- New Zealand (2):
  - Pfizer Investigational Site, Hamilton, Waikato Region
  - Pfizer Investigational Site, Auckland
- Norway (14):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Bodø
  - Pfizer Investigational Site, Fredrikstad
  - Pfizer Investigational Site, Haugesund
  - Pfizer Investigational Site, Levanger
  - Pfizer Investigational Site, Mo i Rana
  - Pfizer Investigational Site, Molde
  - Pfizer Investigational Site, Notodden
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Rissa
  - Pfizer Investigational Site, Rjukan
  - Pfizer Investigational Site, Sandefjord
  - Pfizer Investigational Site, Tromsø
  - Pfizer Investigational Site, Tønsberg
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Poland (8):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Gliwice
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Opole
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Sopot
  - Pfizer Investigational Site, Warsaw
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Evora
- Romania (3):
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Cluj-Napoca
  - Pfizer Investigational Site, Timișoara
- Pfizer Investigational Site, Saint Petersburg, Russia
- Serbia (2):
  - Pfizer Investigational Site, Kamenitz, Serbia
  - Pfizer Investigational Site, Belgrade
- Slovakia (3):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
- Pfizer Investigational Site, Ljubljana, Slovenia
- South Africa (2):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Observatory
- Spain (17):
  - Pfizer Investigational Site, Albacete, Albacete
  - Pfizer Investigational Site, Alcoy, Alicante
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Sant Joan d'Alacant, Alicante
  - Pfizer Investigational Site, Badajoz, Badajoz
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Guadalajara, Guadalajara
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Barbastro, Huesca
  - Pfizer Investigational Site, Lleida, Lleida
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Reus, Tarragona
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Zaragoza, Zaragoza
- Sweden (16):
  - Pfizer Investigational Site, Borås, Sweden
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Halmstad
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Kristianstad
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Motala
  - Pfizer Investigational Site, Nässjö
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, Vaxjo
  - Pfizer Investigational Site, Värnamo
  - Pfizer Investigational Site, Västerås
  - Pfizer Investigational Site, Västervik
- Switzerland (4):
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bellinzona
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Geneva
- United Kingdom (35):
  - Pfizer Investigational Site, Huntingdon, Cambs
  - Pfizer Investigational Site, Bournemouth, Dorset
  - Pfizer Investigational Site, Hull, East Yorkshire
  - Pfizer Investigational Site, Epping, Essex
  - Pfizer Investigational Site, Westcliff-on-Sea, Essex
  - Pfizer Investigational Site, Newport, Gwent
  - Pfizer Investigational Site, Bangor, Gwynedd
  - Pfizer Investigational Site, Salterhebble, Halifax
  - Pfizer Investigational Site, Gosport, Hants
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, Harrogate, N. Yorkshire
  - Pfizer Investigational Site, Londonderry, Northern Ireland
  - Pfizer Investigational Site, Taunton, Somerset
  - Pfizer Investigational Site, Swansea, South Wales
  - Pfizer Investigational Site, York, Yorkshire
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Bradford
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, East Kilbride
  - Pfizer Investigational Site, Huddersfield
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Lincoln
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Luton
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Shrewsbury
  - Pfizer Investigational Site, Somerset
  - Pfizer Investigational Site, Southampton
  - Pfizer Investigational Site, Steeton
  - Pfizer Investigational Site, Stoke-on-Trent
  - Pfizer Investigational Site, Telford
  - Pfizer Investigational Site, Wythenshawe, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=96-OEXE-031&StudyName=Randomized%20Trial%20Of%20Exemestane%20Versus%20Continued%20Tamoxifen%20In%20Postmenopausal%20Women%20With%20Early%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The publication describing study results (Coombes RC et al; N Engl J Med 350; 1119) stated that 4742 participants were enrolled in study. It was later discovered that 2 participants were randomized twice. Hence, 4740 participants were enrolled in this study.
Pre-assignment Details: Main study also included 3 sub-studies only for the purpose of tolerability assessment: endometrial status, bone metabolism and quality of life (QoL). Out of 4740 enrolled participants, data for 16 participants from a center were excluded since it was considered unreliable. Results are reported for remaining 4724 participants.
Groups:
- Exemestane: Participants diagnosed with breast cancer who remained disease-free after previously receiving 2 to 3 years of tamoxifen 20 milligram (mg) or 30 mg tablet-in-capsule orally once daily as per standard medical practice, received exemestane (Aromasin) 25 mg tablet-in-capsule orally once daily for the remainder of 5-year period.
- Tamoxifen: Participants diagnosed with breast cancer who remained disease-free after previously receiving 2 to 3 years of tamoxifen 20 mg or 30 mg tablet-in-capsule orally once daily as per standard medical practice, received the same dose of tamoxifen tablet-in-capsule orally once daily for the remainder of 5-year period.
Period: Overall Study
Arm/Group | Exemestane | Tamoxifen
Started | 2352 | 2372
Treated | 2321 (8 participants randomized to receive exemestane, received tamoxifen. Reported as per randomization.) | 2337 (7 participants randomized to receive tamoxifen, received exemestane. Reported as per randomization.)
Completed | 1810 | 1830
Not Completed | 542 | 542
Not completed — Adverse Event | 170 | 145
Not completed — Withdrawal by Subject | 150 | 107
Not completed — Protocol Violation | 19 | 22
Not completed — Death | 22 | 16
Not completed — Lost to Follow-up | 15 | 10
Not completed — Recurrence | 109 | 179
Not completed — Randomized, but not treated | 31 | 35
Not completed — Other | 26 | 28

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants assigned to the treatment group to which they were randomized, irrespective of the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane | Tamoxifen | Total
Number analyzed (Participants) | 2352 | 2372 | 4724
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.78 (8.12) | 63.69 (8.22) | 63.73 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2352 | 2372 | 4724
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS) at Month 36 Post-Randomization: Main Study
Description: DFS defined as time from randomization to earliest documentation of breast cancer relapse or death from any cause. DFS at Month 36 post-randomization was defined as probability of participants alive and disease-free at 36 months after the randomization. Participants withdrawn from the study for any reason in the absence of relapse were censored at the date they were last seen. Relapse was categorized as follows: loco-regional: ipsilateral breast or axillary nodal relapse; distant: distant relapse, including supraclavicular nodes; second primary breast cancer: contralateral breast cancer, excluding ductal carcinoma in situ.
Time Frame: Baseline up to Month 36
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: probability of DFS
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 2352 | 2372
probability of DFS | 0.90 [0.89 to 0.92] | 0.86 [0.85 to 0.88]
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; Test type: Superiority or Other; p = 0.00003, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.58 to 0.82]

2. Secondary Outcome: Overall Survival (OS) at Month 36 Post-Randomization: Main Study
Description: OS was defined as the duration from randomization to death (due to any cause). OS at Month 36 post-randomization was defined as probability of participants' survival at 36 months after the randomization. For participants who were alive, OS was censored at the last available assessment. Probability of OS at Month 36 post-randomization was reported using Kaplan-Meier estimates at Month 36 post-randomization based on 120-month follow-up data.
Time Frame: Baseline up to Month 120
Population: ITT population included all participants assigned to the treatment group to which they were randomized, irrespective of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: probability of OS
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 2352 | 2372
probability of OS | 0.953 [0.945 to 0.962] | 0.941 [0.932 to 0.951]
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; Test type: Superiority or Other; p = 0.15737, Log Rank; Hazard Ratio (HR) = 0.913, 95% CI 2-sided [0.806 to 1.036]

3. Secondary Outcome: Number of Events of Second Breast Cancer in Contralateral Breast: Main Study
Description: Number of events of second primary breast cancer in contralateral breast (excluding ductal carcinoma in situ) were reported.
Time Frame: Baseline up to Month 120
Population: as for outcome 2
Measure: Number; unit: events
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 2352 | 2372
events | 57 | 75

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine and Proximal Femur (Total Hip) Bone Mineral Density (BMD) at 6, 12, 24 Months On-treatment and 24 Months Post-treatment: Bone Metabolism Sub-study
Description: BMD measurements for Lumbar spine (LS) and Proximal Femur (Total Hip [TH]) were performed using dual energy X-ray absorptiometry (DXA) for participants who entered the bone-metabolism sub-study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 6, 12, 24 months after randomization (on-treatment), 24 months post-treatment
Population: Evaluable population for bone metabolism substudy: all treated participants who did not violate any exclusion criteria, received treatment for at least 9 months and had baseline and at least on-treatment Month 12 and/or Month 24 assessment available for parameter to be analyzed. Participants were analyzed according to treatment actually received.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 84 | 96
percent change
  Change at 6 months on-treatment: LS (n=84,96) | -2.64 (2.89) | -0.22 (2.55)
  Change at 6 months on-treatment: TH (n=82,96) | -1.31 (2.20) | -0.13 (1.90)
  Change at 12 months on-treatment: LS (n=82,96) | -2.98 (3.30) | -0.19 (3.53)
  Change at 12 months on-treatment: TH (n=82,95) | -2.17 (2.34) | -0.39 (2.17)
  Change at 24 months on-treatment: LS (n=82,92) | -3.69 (4.12) | -0.47 (3.38)
  Change at 24 months on-treatment: TH (n=79,93) | -2.81 (2.61) | -0.91 (2.66)
  Change at 24 months post-treatment: LS (n=74,81) | -2.17 (5.09) | -3.44 (4.28)
  Change at 24 months post-treatment: TH (n=73,84) | -3.06 (4.35) | -4.15 (4.01)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 6 months on-treatment (lumbar spine): p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 2.43, 95% CI 2-sided [1.63 to 3.23]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months on-treatment (total hip): p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [0.57 to 1.79]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 12 months on-treatment (lumbar spine): p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 2.79, 95% CI 2-sided [1.77 to 3.81]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months on-treatment (total hip): p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [1.12 to 2.46]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 24 months on-treatment (lumbar spine): p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 3.22, 95% CI 2-sided [2.10 to 4.35]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months on-treatment (total hip): p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 1.90, 95% CI 2-sided [1.10 to 2.69]

5. Secondary Outcome: Percent Change From Baseline in Femoral Neck and Femoral Wards Bone Mineral Density (BMD) at 6, 12 and 24 Months On-treatment and 24 Months Post-treatment: Bone Metabolism Sub-study
Description: BMD measurements for femoral neck (FN) and femoral wards (FW) were performed using dual energy X-ray absorptiometry (DXA) for participants who entered the bone-metabolism sub-study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 6, 12, 24 months after randomization (on-treatment), 24 months post-treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 82 | 95
percent change
  Change at 6 months on-treatment: FN (n=82,94) | -1.91 (3.17) | -0.30 (3.75)
  Change at 6 months on-treatment: FW (n=82,94) | -2.02 (4.57) | 0.32 (5.53)
  Change at 12 months on-treatment: FN (n=82,95) | -2.56 (3.26) | -0.32 (3.60)
  Change at 12 months on-treatment: FW (n=81,95) | -3.51 (4.88) | -1.30 (5.84)
  Change at 24 months on-treatment: FN (n=78,89) | -4.00 (3.61) | -0.78 (4.85)
  Change at 24 months on-treatment: FW (n=72,87) | -4.75 (6.29) | -1.86 (7.32)
  Change at 24 months post-treatment: FN (n=61,69) | -4.10 (5.57) | -4.95 (6.46)
  Change at 24 months post-treatment: FW (n=60,68) | -6.07 (7.63) | -8.60 (8.15)

6. Secondary Outcome: Change From Baseline in Lumbar Spine and Proximal Femur (Total Hip) Bone Mineral Density (BMD) T-scores at 6, 12 and 24 Months On-treatment and 24 Months Post-treatment: Bone Metabolism Sub-study
Description: BMD measurements for Lumbar spine (LS) and Proximal Femur (Total Hip [TH]) were performed using dual energy X-ray absorptiometry (DXA) for participants who entered the bone-metabolism sub-study. Results were scored as T-score. T-score indicated how many standard deviations higher or lower participant's value was when compared to the young normal reference mean. Using the World Health Organization (WHO) criteria for osteoporosis, a T-score of greater than or equal to (>=)-1.0 was classified as normal, a T-score of greater than -2.5 to less than -1.0 as osteopenic, and a T-score less than or equal to (<=)-2.5 as osteoporotic. Here 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 6, 12, 24 months after randomization (on-treatment), 24 months post-treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 86 | 99
T-score
  Baseline: LS (n=86,99) | -0.62 (1.12) | -0.45 (1.14)
  Baseline: TH (n=86,99) | -0.27 (0.97) | -0.12 (1.01)
  Change at 6 months on-treatment: LS (n=84,96) | -0.24 (0.26) | -0.02 (0.23)
  Change at 6 months on-treatment: TH (n=82,96) | -0.10 (0.19) | -0.00 (0.16)
  Change at 12 months on-treatment: LS (n=82,96) | -0.26 (0.30) | -0.02 (0.32)
  Change at 12 months on-treatment: TH (n=82,95) | -0.16 (0.21) | -0.03 (0.18)
  Change at 24 months on-treatment: LS (n=82,92) | -0.32 (0.41) | -0.04 (0.31)
  Change at 24 months on-treatment: TH (n=79,93) | -0.21 (0.27) | -0.07 (0.24)
  Change at 24 months post-treatment: LS (n=74,81) | -0.21 (0.47) | -0.33 (0.41)
  Change at 24 months post-treatment: TH (n=73,84) | -0.25 (0.38) | -0.34 (0.33)

7. Secondary Outcome: Percentage of Bone Specific Alkaline Phosphatase (BAP) Serum Concentration Relative to Baseline: Bone Metabolism Sub-study
Description: Bone specific alkaline phosphatase (BAP) serum concentration analyzed using enzyme immuno assay (EIA) at post-baseline time points was expressed as percentage of baseline BAP serum concentration. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30 months after randomization (on-treatment), 36 months after randomization (end of treatment), 12, 24 months post-treatment
Population: As treated population for bone metabolism sub-study included all treated participants, irrespective of the treatment duration and allocated to the group that corresponded to the treatment they actually received. Analysis population for biomarkers included as treated population with baseline and at least 1 on-treatment assessment available.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline concentration
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 83 | 96
percentage of baseline concentration
  3 months: on-treatment (n=81, 92) | 113.47 [108.74 to 118.41] | 104.35 [100.03 to 108.85]
  6 months: on-treatment (n=83, 95) | 121.01 [107.99 to 135.60] | 104.34 [99.18 to 109.76]
  9 months: on-treatment (n=79, 92) | 139.62 [131.65 to 148.06] | 98.17 [92.95 to 103.67]
  12 months: on-treatment (n=82, 96) | 148.96 [139.83 to 158.68] | 100.47 [94.36 to 106.97]
  18 months: on-treatment (n=80, 95) | 158.33 [147.97 to 169.41] | 102.72 [96.18 to 109.69]
  24 months: on-treatment (n=81, 90) | 155.89 [145.04 to 167.56] | 105.12 [98.36 to 112.35]
  30 months: on-treatment (n=50, 65) | 144.89 [125.83 to 166.83] | 108.33 [99.51 to 117.94]
  36 months: end of treatment (n=19, 31) | 150.82 [127.82 to 177.97] | 113.87 [101.28 to 128.03]
  12 months: post-treatment (n=67, 87) | 140.19 [129.98 to 151.19] | 149.69 [138.34 to 161.97]
  24 months: post-treatment (n=62, 77) | 128.73 [114.70 to 144.48] | 142.20 [129.09 to 156.64]

8. Secondary Outcome: Percentage of C-Terminal Telopeptide (CTX) Serum Concentration Relative to Baseline: Bone Metabolism Sub-study
Description: C-terminal telopeptide (CTX) serum concentration analyzed using competitive enzyme-linked immunosorbent assay (ELISA) at post-baseline time points was expressed as percentage of baseline CTX serum concentration. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline concentration
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 83 | 96
percentage of baseline concentration
  3 months: on-treatment (n=81, 93) | 144.14 [127.25 to 163.27] | 99.19 [89.37 to 110.09]
  6 months: on-treatment (n=83, 95) | 197.47 [176.51 to 220.92] | 93.67 [84.75 to 103.51]
  9 months: on-treatment (n=79, 92) | 226.04 [202.51 to 252.30] | 94.40 [85.44 to 104.29]
  12 months: on-treatment (n=81, 96) | 232.69 [206.42 to 262.31] | 94.59 [86.27 to 103.71]
  18 months: on-treatment (n=80, 95) | 199.68 [171.75 to 232.15] | 90.35 [81.82 to 99.76]
  24 months: on-treatment (n=81, 90) | 177.80 [154.58 to 204.50] | 88.80 [78.96 to 99.87]
  30 months: on-treatment (n=50, 65) | 179.29 [150.83 to 213.11] | 91.62 [80.20 to 104.66]
  36 months: end of treatment (n=19, 31) | 130.00 [94.91 to 178.06] | 99.34 [81.16 to 121.58]
  12 months: post-treatment (n=67, 87) | 110.87 [94.93 to 129.49] | 136.50 [121.05 to 153.91]
  24 months: post-treatment (n=62, 77) | 100.34 [84.62 to 118.98] | 124.03 [109.98 to 139.88]

9. Secondary Outcome: Percentage of Osteocalcin (OC) and Procollagen T1 C-Peptide (PICP) Serum Concentration Relative to Baseline: Bone Metabolism Sub-study
Description: Osteocalcin (OC) serum concentration analyzed using ELISA and procollagen T1 c-peptide (PICP) serum concentration analyzed using sandwich EIA at post-baseline time points was expressed as percentage of baseline OC serum concentration and baseline PICP serum concentration, respectively. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points, for each group respectively.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline concentration
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 83 | 96
percentage of baseline concentration
  3 months, on-treatment: OC (n=81, 92) | 149.49 [137.88 to 162.09] | 101.02 [94.14 to 108.40]
  3 months, on-treatment: PICP (n=81, 92) | 117.23 [109.63 to 125.35] | 102.19 [97.34 to 107.27]
  6 months, on-treatment: OC (n=83, 95) | 193.44 [177.49 to 210.81] | 97.69 [91.78 to 103.98]
  6 months, on-treatment: PICP (n=83, 95) | 133.50 [125.30 to 142.23] | 99.78 [95.18 to 104.61]
  9 months, on-treatment: OC (n=79, 93) | 230.41 [209.80 to 253.05] | 92.52 [86.02 to 99.50]
  9 months, on-treatment: PICP (n=79, 92) | 131.73 [124.27 to 139.63] | 96.52 [91.21 to 102.14]
  12 months, on-treatment: OC (n=82, 96) | 227.59 [208.40 to 248.56] | 95.75 [88.46 to 103.65]
  12 months, on-treatment: PICP (n=82, 96) | 128.68 [122.22 to 135.50] | 100.18 [95.23 to 105.39]
  18 months, on-treatment: OC (n=80, 95) | 230.72 [207.16 to 256.95] | 93.98 [87.54 to 100.90]
  18 months, on-treatment: PICP (n=80, 95) | 125.40 [116.86 to 134.56] | 103.25 [97.38 to 109.47]
  24 months, on-treatment: OC (n=81, 90) | 190.18 [171.07 to 211.41] | 89.29 [82.19 to 97.00]
  24 months: on-treatment: PICP (n=81, 90) | 123.75 [115.11 to 133.05] | 103.94 [97.75 to 110.52]
  30 months, on-treatment: OC (n=50, 65) | 187.23 [165.02 to 212.43] | 87.34 [79.64 to 95.79]
  30 months, on-treatment: PICP (n=50, 65) | 113.76 [102.05 to 126.82] | 103.36 [94.57 to 112.97]
  36 months, end of treatment: OC (n=19, 30) | 167.03 [121.37 to 229.86] | 90.77 [76.63 to 107.52]
  36 months, end of treatment: PICP (n=19, 31) | 95.33 [79.82 to 113.84] | 87.22 [76.34 to 99.66]
  12 months, post-treatment: OC (n=67, 87) | 143.85 [125.83 to 164.44] | 152.32 [135.49 to 171.24]
  12 months, post-treatment: PICP (n=67, 87) | 91.53 [84.27 to 99.42] | 108.67 [100.59 to 117.39]
  24 months, post-treatment: OC (n=62, 77) | 130.78 [114.03 to 150.00] | 146.36 [128.87 to 166.22]
  24 months, post-treatment: PICP (n=62, 77) | 90.46 [81.68 to 100.19] | 100.74 [92.95 to 109.19]

10. Secondary Outcome: Percentage of Deoxy-pyridinoline (DPD) Urine Concentration Relative to Baseline: Bone Metabolism Sub-study
Description: Deoxy-pyridinoline (DPD) urine concentration (adjusted for urinary creatinine) analyzed using competitive EIA at post-baseline time points was expressed as percentage of baseline DPD urine concentration. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline concentration
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 83 | 97
percentage of baseline concentration
  3 months: on-treatment (n=82, 91) | 130.49 [121.56 to 140.07] | 106.99 [99.66 to 114.85]
  6 months: on-treatment (n=83, 95) | 145.13 [133.61 to 157.64] | 103.42 [96.64 to 110.68]
  9 months: on-treatment (n=80, 92) | 160.12 [147.40 to 173.93] | 101.08 [94.85 to 107.72]
  12 months: on-treatment (n=82, 97) | 155.53 [143.40 to 168.70] | 104.51 [98.23 to 111.19]
  18 months: on-treatment (n=77, 96) | 139.57 [129.65 to 150.25] | 99.25 [93.11 to 105.78]
  24 months: on-treatment (n=78, 90) | 135.30 [125.10 to 146.33] | 99.11 [92.56 to 106.12]
  30 months: on-treatment (n=49, 63) | 121.39 [108.66 to 135.62] | 95.97 [87.65 to 105.07]
  36 months: end of treatment (n=19, 31) | 107.64 [89.11 to 130.02] | 101.04 [86.77 to 117.65]
  12 months: post-treatment (n=65, 84) | 117.94 [107.07 to 129.92] | 128.47 [118.34 to 139.46]
  24 months: post-treatment (n=61, 77) | 105.50 [96.08 to 115.84] | 120.84 [112.37 to 129.96]

11. Secondary Outcome: Percentage of N-telopeptide of Type 1 Collagen (NTX) Urine Concentration Relative to Baseline: Bone Metabolism Sub-study
Description: N-telopeptide of Type 1 collagen (NTX) urine concentration (adjusted for urinary creatinine) analyzed using competitive inhibition EIA at post-baseline time points was expressed as percentage of baseline NTX urine concentration. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline concentration
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 83 | 97
percentage of baseline concentration
  3 months: on-treatment (n=82, 91) | 128.35 [118.11 to 139.48] | 101.92 [94.39 to 110.05]
  6 months: on-treatment (n=83, 95) | 153.67 [141.89 to 166.44] | 100.64 [92.92 to 109.00]
  9 months: on-treatment (n=80, 92) | 168.15 [152.93 to 184.90] | 101.44 [92.13 to 111.68]
  12 months: on-treatment (n=82, 97) | 177.58 [160.20 to 196.85] | 104.42 [96.57 to 112.91]
  18 months: on-treatment (n=77, 96) | 171.46 [153.32 to 191.75] | 98.74 [89.88 to 108.46]
  24 months: on-treatment (n=78, 90) | 167.87 [148.36 to 189.95] | 104.55 [93.40 to 117.03]
  30 months: on-treatment (n=49, 63) | 168.52 [144.54 to 196.48] | 96.51 [83.74 to 111.22]
  36 months: end of treatment (n=19, 31) | 152.13 [112.43 to 205.87] | 105.58 [84.56 to 131.83]
  12 months: post-treatment (n=65, 84) | 121.00 [101.05 to 144.88] | 158.12 [139.47 to 179.26]
  24 months: post-treatment (n=61, 77) | 108.18 [108.18 to 129.77] | 143.98 [124.26 to 166.83]

12. Secondary Outcome: Number of Participants With Fracture: Bone Metabolism Sub-study
Time Frame: Baseline up to 24 months post-treatment
Population: As treated population for bone metabolism sub-study included all treated participants, irrespective of the treatment duration and allocated to the group that corresponded to the treatment they actually received.
Measure: Number; unit: participants
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 101 | 105
participants | 7 | 10

13. Secondary Outcome: Change From Baseline in Treatment Outcome Index (TOI) at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The TOI was defined as the sum of 23 items based on following Functional Assessment of Cancer Therapy - Breast version [FACT-B] subscales: Physical well-being (7 items), Functional well-being (7 items), Breast cancer subscale (9 items). Each item was scaled from 0='Not at all' to 4='Very much'. Total TOI score ranged from 0 to 92, where higher TOI score indicated better health-related quality of life (QoL). A change of five points in the TOI scores was considered clinically meaningful. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively. Results for 30, 36, 48, 60 months were not reported because data for these time points was only summarized as graphical presentation.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: ITT population for QoL sub-study included all randomized participants with available data for any given endpoint and were grouped according to randomized treatment, irrespective of whether they were actually treated or not.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 251 | 251
units on a scale
  Change at 3 months (n=251, 251) | -0.61 (7.72) | -0.16 (7.24)
  Change at 6 months (n=244, 243) | -2.10 (9.66) | -0.01 (7.96)
  Change at 9 months (n=242, 235) | -1.18 (8.62) | 0.17 (8.10)
  Change at 12 months (n=230, 238) | -0.40 (8.03) | -0.66 (8.49)
  Change at 18 months (n=232, 227) | -0.95 (8.99) | -0.11 (8.32)
  Change at 24 months (n=221, 213) | -0.57 (9.06) | 0.54 (8.36)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.500, t-test, 2 sided; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.76 to 0.86]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-3.67 to -0.52]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.079, t-test, 2 sided; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-2.86 to 0.16]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.729, t-test, 2 sided; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-1.24 to 1.77]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.302, t-test, 2 sided; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-2.43 to 0.75]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.187, t-test, 2 sided; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-2.76 to 0.54]

14. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Endocrine Subscale (FACT-ES) Total Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The FACT-ES assessed health-related QoL in participants with breast cancer. ES subscale comprised of 18 items (hot flushes,cold sweats,night sweats, vaginal discharge,vaginal irritation,vaginal bleeding,vaginal dryness,discomfort with intercourse,lost interest in sex,gained weight,light headed/dizzy,vomiting,had diarrhea,headaches,felt bloated,breast tenderness,mood swings, felt irritable).Participants indicated how true a statement was for them using a 5-point scale from 0 (not at all) to 4 (very much). For items that were negatively framed, the scores were reversed for the analysis so that higher scores equated to a good QoL. Total FACT-ES score was calculated as sum of all the 18 items and ranged from 0 to 72, where higher score indicated better QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: ITT population for QoL sub-study. Results for 30, 36, 48, 60 months were not reported because data for these time points was only summarized as graphical presentation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 254 | 253
units on a scale
  Change at 3 months (n=254, 253) | 0.04 (6.67) | 0.70 (6.40)
  Change at 6 months (n=245, 243) | 0.17 (7.26) | 0.96 (6.54)
  Change at 9 months (n=243, 238) | 1.10 (6.54) | 1.32 (6.29)
  Change at 12 months (n=233, 236) | 1.98 (6.72) | 1.15 (7.08)
  Change at 18 months (n=235, 226) | 1.25 (7.52) | 1.41 (6.67)
  Change at 24 months (n=222, 214) | 1.93 (7.26) | 1.51 (6.87)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.260, t-test, 2 sided; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.80 to 0.49]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.209, t-test, 2 sided; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-2.02 to 0.44]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.698, t-test, 2 sided; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.38 to 0.92]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.192, t-test, 2 sided; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.42 to 2.09]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.813, t-test, 2 sided; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-1.46 to 1.15]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.537, t-test, 2 sided; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.91 to 1.75]

15. Secondary Outcome: Change From Baseline in Total Functional Assessment of Cancer Therapy - General Breast and Endocrine (FACT-GBE) Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: FACT-GBE assessed health-related quality of life (QoL) in participants with breast cancer. It consisted of 56 items,summarized to 7 subscales(subscale 1 to 6 constituted total FACT-B and subscale 7 constituted total ES):physical well-being(7 items), social/family well-being(7 items),relationship with doctor (2 items),emotional well-being(6 items),functional well-being(7 items),breast cancer subscale(9 items),endocrine symptoms(18 items). Participants indicated how true a statement had been for them using 5-point scale from 0(not at all) to 4(very much). For items that were negatively framed,scores were reversed for analysis so that higher scores equated to good QoL. Total FACT-GBE score=sum of all 56 items(range 0 to 224, where higher score indicated better QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 252 | 252
units on a scale
  Change at 3 months (n=252, 252) | -0.91 (17.41) | -0.38 (16.17)
  Change at 6 months (n=244, 243) | -3.12 (17.84) | -0.04 (16.21)
  Change at 9 months (n=243, 236) | -1.28 (15.09) | -0.38 (17.99)
  Change at 12 months (n=229, 236) | 0.38 (18.91) | -0.53 (14.71)
  Change at 18 months (n=232, 225) | -0.67 (17.37) | 0.06 (16.26)
  Change at 24 months (n=220, 212) | -1.48 (22.44) | 1.43 (16.32)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.727, t-test, 2 sided; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-3.46 to 2.42]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.047, t-test, 2 sided; Mean Difference (Final Values) = -3.08, 95% CI 2-sided [-6.12 to -0.05]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.553, t-test, 2 sided; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-3.88 to 2.08]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.563, t-test, 2 sided; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-2.17 to 3.99]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.643, t-test, 2 sided; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-3.83 to 2.36]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.126, t-test, 2 sided; Mean Difference (Final Values) = -2.91, 95% CI 2-sided [-6.63 to 0.82]

16. Secondary Outcome: Change From Baseline in Physical Well-Being (PWB) Subscale Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The PWB subscale assessed physical well-being related QoL in participants with breast cancer. PWB subscale comprised of 7 items (energy lack, nausea, family needs, pain, side effects, felt ill, forced to stay in bed). Participants indicated how true a statement had been for them using a 5-point scale from 0 (not at all) to 4 (very much). For items that were negatively framed, the scores were reversed for the analysis so that higher scores equated to a good QoL. Total PWB score was calculated as the sum of all the 7 items and ranged from 0 to 28, where higher score indicated better physical well-being related QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 253 | 252
units on a scale
  Change at 3 months (n=253, 252) | -0.32 (3.05) | -0.02 (2.98)
  Change at 6 months(n=246, 244) | -1.08 (4.16) | 0.13 (2.88)
  Change at 9 months (n=242, 237) | -0.37 (3.16) | 0.06 (3.16)
  Change at 12 months (n=233, 238) | -0.26 (2.90) | -0.12 (3.30)
  Change at 18 months(n=234, 228) | -0.19 (3.09) | 0.02 (2.81)
  Change at 24 months (n=223, 214) | -0.005 (0.208) | 0.22 (0.214)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.265, t-test, 2 sided; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.83 to 0.23]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-1.84 to -0.57]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.132, t-test, 2 sided; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.00 to 0.13]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.635, t-test, 2 sided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.70 to 0.43]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.449, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.75 to 0.33]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.454, t-test, 2 sided; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.81 to 0.36]

17. Secondary Outcome: Change From Baseline in Social/Family Well-Being (SWB) Sub-scale Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The SWB subscale assessed social/family well-being related QoL in participants with breast cancer. SWB subscale comprised of 7 items (distant from friends, emotional support, support from friends, family acceptance, family communication, close to main support, sexual satisfaction). Participants indicated how true a statement had been for them using a 5-point scale from 0 (not at all) to 4 (very much). For items that were negatively framed, the scores were reversed for the analysis so that higher scores equated to a good QoL. Total SWB score was calculated as the sum of all the 7 items and ranged from 0 to 28, where higher score indicated better social/family well-being related QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 252 | 249
units on a scale
  Change at 3 months (n=252, 249) | -0.25 (3.90) | -0.37 (3.59)
  Change at 6 months (n=245, 241) | -0.43 (3.84) | -0.47 (4.01)
  Change at 9 months (n=242, 235) | -0.58 (3.61) | -0.53 (4.22)
  Change at 12 months (n=231, 235) | 0.05 (4.03) | -0.56 (3.87)
  Change at 18 months(n=234, 226) | -0.5 (3.62) | -0.69 (4.31)
  Change at 24 months (n=219, 212) | -0.99 (4.96) | -0.72 (4.44)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.712, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.53 to 0.335]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.899, t-test, 2 sided; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.65 to 0.356]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.882, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.76 to 0.359]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.604, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.54 to 0.37]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.562, t-test, 2 sided; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.16 to 0.454]

18. Secondary Outcome: Change From Baseline in Relationship With Doctor (RWD) Subscale Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Substudy
Description: The RWD subscale assessed relationship with doctor in participants with breast cancer. RWD subscale comprised of 2 items (confidence in doctors, doctor answered questions). Participants indicated how true a statement had been for them using a 5-point scale from 0 (not at all) to 4 (very much). Total RWD score was calculated as the sum of the 2 items and ranged from 0 to 8, where higher score indicated better relationship with doctor. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 254 | 250
units on a scale
  Change at 3 months (n=254, 250) | 0.07 (1.20) | 0.08 (0.94)
  Change at 6 months (n=244, 240) | -0.02 (1.34) | -0.04 (1.14)
  Change at 9 months (n=243, 235) | -0.06 (1.12) | -0.07 (1.06)
  Change at 12 months (n=233, 233) | -0.01 (1.20) | -0.07 (1.12)
  Change at 18 months (n=233, 222) | -0.03 (1.27) | -0.21 (1.20)
  Change at 24 months (n=221, 213) | -0.005 (1.25) | -0.12 (1.14)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.892, t-test, 2 sided; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.20 to 0.18]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.881, t-test, 2 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.21 to 0.24]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.883, t-test, 2 sided; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.18 to 0.21]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.604, t-test, 2 sided; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.16 to 0.27]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.118, t-test, 2 sided; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.05 to 0.41]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.307, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.11 to 0.34]

19. Secondary Outcome: Change From Baseline in Emotional Well-Being (EWB) Subscale Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The EWB subscale assessed emotional well-being related QoL in participants with breast cancer. EWB subscale comprised of 6 items (felt sad, proud of coping, lost hope, felt nervous, worried about dying, worried about condition worsening). Participants indicated how true a statement had been for them using a 5-point scale from 0 (not at all) to 4 (very much). For items that were negatively framed, the scores were reversed for the analysis so that higher scores equate to a good QoL. Total EWB score was calculated as the sum of the 6 items and ranged from 0 to 24, where higher score indicated better emotional well-being related QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 255 | 252
units on a scale
  Change at 3 months (n=255, 252) | 0.06 (2.84) | -0.01 (2.77)
  Change at 6 months (n=246, 243) | -0.32 (2.88) | -0.1 (3.10)
  Change at 9 months (n=243, 236) | -0.47 (3.05) | -0.27 (3.12)
  Change at 12 months (n=232, 235) | -0.03 (2.55) | -0.33 (2.86)
  Change at 18 months (n=235, 226) | -0.3 (3.05) | -0.04 (3.26)
  Change at 24 months (n=222, 214) | -0.18 (3.05) | 0.07 (3.09)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.792, t-test, 2 sided; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.42 to 0.56]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.405, t-test, 2 sided; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.76 to 0.31]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.484, t-test, 2 sided; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.75 to 0.36]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.229, t-test, 2 sided; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.19 to 0.80]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.381, t-test, 2 sided; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.84 to 0.32]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.405, t-test, 2 sided; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.82 to 0.33]

20. Secondary Outcome: Change From Baseline in Functional Well-Being (FWB) Sub-scale Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The FWB subscale assessed functional well-being related QoL in participants with breast cancer. FWB subscale comprised of 7 items (able to work, work fulfilled, able to enjoy life, acceptance of illness, sleeping well, enjoyed normal fun activities, contented with QoL). Participants indicated how true a statement had been for them using a 5-point scale from 0 (not at all) to 4 (very much). Total FWB score was calculated as the sum of the 7 items and ranged from 0 to 28, where higher score indicated better functional well-being related QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 254 | 253
units on a scale
  Change at 3 months (n=254, 253) | -0.32 (3.79) | -0.18 (3.32)
  Change at 6 months (n=246, 244) | -0.77 (4.31) | -0.43 (4.01)
  Change at 9 months (n=243, 238) | -1.03 (3.96) | -0.38 (3.62)
  Change at 12 months (n=232, 238) | -0.68 (4.07) | -0.91 (4.38)
  Change at 18 months (n=232, 227) | -0.83 (4.14) | -0.8 (3.89)
  Change at 24 months (n=222, 214) | -0.91 (4.49) | -0.45 (3.72)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.648, t-test, 2 sided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.77 to 0.48]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.366, t-test, 2 sided; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.08 to 0.40]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.062, t-test, 2 sided; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.33 to 0.03]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.545, t-test, 2 sided; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.53 to 1.00]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.932, t-test, 2 sided; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.77 to 0.70]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.244, t-test, 2 sided; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.24 to 0.32]

21. Secondary Outcome: Change From Baseline in Breast Cancer Subscale (BCS) Score at 3, 6, 9, 12, 18, 24, 30, 36, 48 and 60 Months: QoL Sub-study
Description: The BCS subscale assessed health related QoL in participants with breast cancer. BCS subscale comprised of 9 items (short of breath, self-conscious dress, tender/swollen arms, sexually attractive, bothered by hair loss, worried about familial risk, worried about family stress, bothered by weight change, able to feel like a woman). Participants indicated how true a statement had been for them using a 5-point scale from 0 (not at all) to 4 (very much). For items that were negatively framed, the scores were reversed for the analysis so that higher scores equated to a good QoL. Total BCS score was calculated as the sum of the 9 items and ranged from 0 to 36, where higher score indicated better QoL. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 3, 6, 9, 12, 18, 24, 30, 36, 48, 60 months after randomization
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 255 | 252
units on a scale
  Change at 3 months (n=255, 252) | 0.05 (3.76) | -0.003 (3.96)
  Change at 6 months (n=246, 244) | -0.33 (4.17) | 0.17 (4.31)
  Change at 9 months (n=243, 239) | 0.3 (3.99) | 0.48 (4.22)
  Change at 12 months (n=233, 238) | 0.61 (4.08) | 0.38 (4.12)
  Change at 18 months (n=233, 227) | 0.06 (4.61) | 0.67 (4.35)
  Change at 24 months (n=222, 214) | 0.36 (4.33) | 0.72 (4.35)
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 3 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.876, t-test, 2 sided; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.62 to 0.73]
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 6 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.195, t-test, 2 sided; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.25 to 0.26]
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 9 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.630, t-test, 2 sided; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.92 to 0.55]
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.530, t-test, 2 sided; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.50 to 0.98]
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 18 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.147, t-test, 2 sided; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.43 to 0.21]
Statistical Analysis 6: Comparison: Exemestane vs Tamoxifen; 24 months: p-value was estimated using 2-sided t-test; Test type: Superiority or Other; p = 0.389, t-test, 2 sided; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.18 to 0.46]

22. Secondary Outcome: Number of Participants With Severe Endocrine Symptoms: QoL Sub-study
Description: Participants indicated prevalence of an endocrine subscale items using a 5-point scale, where 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit), 4 (very much). Endocrine items were grouped in five categories vasomotor (hot flushes, cold sweats, night sweats, sleeping difficulties), neuropsychological (lack of energy, nervous feeling, lightheaded/dizzy, headaches, mood swings, feeling irritable), gastrointestinal symptoms (nausea, gained weight, vomiting, diarrhea, bloated feeling), gynecological symptoms (vaginal discharge, vaginal irritation, vaginal bleeding, vaginal dryness, discomfort with intercourse, lost interest in sex, breast tenderness) and other symptoms (pain, feeling ill, side effects). Number of participants who reported severe endocrine symptoms (defined as response categories "quite a bit" and "very much") were presented.
Time Frame: Baseline up to 24 months after randomization
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 289 | 293
participants
  Hot flushes | 151 | 146
  Cold sweats | 60 | 52
  Night sweats | 115 | 117
  Sleeping difficulties | 110 | 110
  Lack of energy | 115 | 108
  Nervous feeling | 68 | 65
  Lightheaded/dizzy | 34 | 37
  Headaches | 56 | 49
  Mood swings | 70 | 66
  Feeling irritable | 53 | 48
  Nausea | 16 | 14
  Gained weight | 150 | 152
  Vomiting | 6 | 6
  Diarrhea | 20 | 21
  Bloated feeling | 75 | 88
  Vaginal discharge | 36 | 55
  Vaginal irritation | 37 | 45
  Vaginal bleeding | 10 | 11
  Vaginal dryness | 78 | 88
  Discomfort with intercourse | 47 | 45
  Lost interest in sex | 128 | 142
  Breast tenderness | 66 | 76
  Pain | 66 | 60
  Feeling ill | 24 | 24
  Side effects | 54 | 57

23. Secondary Outcome: Percentage of Participants With Endometrial Thickness Greater Than or Equal to (>=) 5 Millimeter (mm): Endometrial Sub-study
Description: Endometrial thickness was assessed using transvaginal ultrasound examination. 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: 6, 12, 24, 36 months after randomization, 6, 12, 24 months post-treatment
Population: Evaluable population for endometrial sub-study included all treated participants who did not violate any exclusion criteria, received treatment for at least 2 years, and had on-treatment endometrial ultrasound examination performed between 22 and 26 months from treatment start. Analysis was based on actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 61 | 52
percentage of participants
  6 months (n=58, 49) | 46.6 | 69.4
  12 months (n=60, 52) | 30.0 | 55.8
  24 months (n=61, 52) | 36.1 | 63.5
  36 months (n=32, 17) | 21.9 | 76.5
  6 months post-treatment (n=16, 17) | 31.3 | 70.6
  12 months post-treatment (n=50, 37) | 30.0 | 32.4
  24 months post-treatment (n=41, 31) | 34.1 | 29.0
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen; 6 months: p-value for percentage of participants with an endometrial thickness of >=5 mm was analyzed using Chi-squared test; Test type: Superiority or Other; p = 0.0174, Chi-squared
Statistical Analysis 2: Comparison: Exemestane vs Tamoxifen; 12 months: p-value for percentage of participants with an endometrial thickness of >=5 mm was analyzed using Chi-squared test; Test type: Superiority or Other; p = 0.0059, Chi-squared
Statistical Analysis 3: Comparison: Exemestane vs Tamoxifen; 24 months: p-value for percentage of participants with an endometrial thickness of >=5 mm was analyzed using Chi-squared test; Test type: Superiority or Other; p = 0.0037, Chi-squared
Statistical Analysis 4: Comparison: Exemestane vs Tamoxifen; 12 months post-treatment: p-value for percentage of participants with an endometrial thickness of >=5 mm was analyzed using Chi-squared test; Test type: Superiority or Other; p = 0.8084, Chi-squared
Statistical Analysis 5: Comparison: Exemestane vs Tamoxifen; 24 months post-treatment: p-value for percentage of participants with an endometrial thickness of >=5 mm was analyzed using Chi-squared test; Test type: Superiority or Other; p = 0.6449, Chi-squared

24. Secondary Outcome: Endometrial Thickness: Endometrial Sub-study
Description: Endometrial thickness was assessed using transvaginal ultrasound examination. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: Baseline, 6, 12, 24, 36 months after randomization, 6, 12, 24 months post-treatment
Population: as for outcome 23
Measure: Median (Full Range); unit: mm
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 60 | 52
mm
  Baseline (n=60, 52) | 6.0 [1.0 to 29.0] | 6.0 [1.0 to 29.0]
  6 months (n=58, 49) | 4.0 [1.0 to 16.0] | 5.9 [2.0 to 23.0]
  12 months (n=59, 52) | 3.3 [1.0 to 20.4] | 5.5 [2.0 to 39.0]
  24 months (n=60, 52) | 4.0 [1.0 to 19.0] | 5.0 [1.0 to 26.0]
  36 months (n=31, 17) | 3.0 [1.0 to 12.0] | 7.0 [2.0 to 24.0]
  6 months post-treatment (n=16, 17) | 3.0 [1.0 to 16.6] | 5.8 [4.0 to 17.0]
  12 months post-treatment (n=49, 37) | 3.0 [1.0 to 17.0] | 4.0 [1.0 to 16.0]
  24 months post-treatment (n=40, 31) | 3.0 [1.0 to 21.0] | 3.8 [1.0 to 10.0]

25. Secondary Outcome: Uterine and Overall Ovary Volume: Endometrial Sub-study
Description: Uterine volume (UV) and ovarian volume was estimated using ultrasonography. Uterine volume = (longitudinal diameter * transverse diameter * anteroposterior diameter of uterus)/(2*1000). Ovary volume = [(longitudinal diameter * transverse diameter * anteroposterior diameter of ovary) * 3.14]/(6*1000). Overall ovary volume (OV) is calculated as the sum of the right and left ovary volume. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome and 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Time Frame: 6, 12, 24, 36 months after randomization, 6, 12, 24 months post-treatment
Population: as for outcome 23
Measure: Median (Full Range); unit: cubic centimeter (cm^3)
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 57 | 51
cubic centimeter (cm^3)
  UV: 6 months (n=57, 47) | 25.2 [5.6 to 180.0] | 36.5 [4.1 to 149.8]
  OV: 6 months (n=8, 6) | 1.8 [1.2 to 9.7] | 1.2 [0.6 to 4.2]
  UV: 12 months (n=56, 49) | 23.3 [0.0 to 58.3] | 39.2 [6.7 to 214.2]
  OV: 12 months (n=6, 5) | 2.3 [1.1 to 6.6] | 2.2 [0.7 to 3.8]
  UV: 24 months (n=54, 51) | 26.3 [6.3 to 73.9] | 40.3 [4.3 to 148.9]
  OV: 24 months (n=5, 6) | 2.0 [0.6 to 4.2] | 2.7 [1.4 to 12.4]
  UV: 36 months (n=30, 18) | 21.5 [4.6 to 116.5] | 36.8 [6.8 to 143.3]
  OV: 36 months (n=3, 2) | 1.5 [0.6 to 2.3] | 2.5 [1.8 to 3.2]
  UV: 6 months post-treatment (n=14, 16) | 25.6 [10.5 to 82.9] | 31.6 [12.9 to 149.5]
  OV: 6 months post-treatment (n=2, 4) | 10.1 [1.4 to 18.7] | 4.7 [2.8 to 11.4]
  UV: 12 months post-treatment (n=42, 35) | 21.7 [8.8 to 96.1] | 30.0 [6.6 to 91.1]
  OV: 12 months post-treatment (n=5, 4) | 2.8 [1.4 to 3.9] | 2.9 [2.1 to 5.3]
  UV: 24 months post-treatment (n=38, 28) | 22.6 [4.8 to 47.2] | 27.8 [7.5 to 71.1]
  OV: 24 months post-treatment (n=4, 4) | 1.6 [1.0 to 3.3] | 3.4 [2.1 to 4.2]

26. Secondary Outcome: Number of Participants With Polyps, Fibroids and Ovarian Cysts: Endometrial Sub-study
Description: Number of participants with presence of polyps (POL) and fibroids (FIB) at post-baseline time points compared to the baseline (BL) status of 'yes', 'no' or 'missing' (that is, participants reporting POL/FIB at post-baseline time points who had yes, no or missing POL/FIB status at baseline, respectively) were presented. Result for number of participants with ovarian cysts was not analyzed at post-baseline time points as very few participants reported ovarian cysts at baseline.
Time Frame: 6, 12, 24, 36 months after randomization, 6, 12, 24 months post-treatment
Population: Evaluable population for endometrial sub-study. Analysis was based on actual treatment received. 'n' signifies those participants who were evaluable for this measure at given time points for each group,respectively.
Measure: Number; unit: participants
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 61 | 52
participants
  FIB: 6 months, BL Yes (n=60,50) | 4 | 6
  FIB: 6 months, BL No (n=60,50) | 2 | 1
  FIB: 6 months, BL Missing (n=60,50) | 2 | 0
  POL: 6 months, BL Yes (n=60,50) | 0 | 0
  POL: 6 months, BL No (n=60,50) | 2 | 0
  POL: 6 months, BL Missing (n=60,50) | 1 | 0
  FIB: 12 months, BL Yes (n=61,52) | 3 | 7
  FIB: 12 months, BL No (n=61,52) | 2 | 1
  FIB: 12 months, BL Missing (n=61,52) | 4 | 1
  POL: 12 months, BL Yes (n=61,52) | 0 | 0
  POL: 12 months, BL No (n=61,52) | 0 | 0
  POL: 12 months, BL Missing (n=61,52) | 1 | 0
  FIB: 24 months, BL Yes (n=61,52) | 3 | 5
  FIB: 24 months, BL No (n=61,52) | 3 | 0
  FIB: 24 months, BL Missing (n=61,52) | 0 | 2
  POL: 24 months, BL Yes (n=61,52) | 1 | 0
  POL: 24 months, BL No (n=61,52) | 0 | 1
  POL: 24 months, BL Missing (n=61,52) | 0 | 0
  FIB: 36 months, BL Yes (n=33,18) | 2 | 1
  FIB: 36 months, BL No (n=33,18) | 3 | 0
  FIB: 36 months, BL Missing (n=33,18) | 0 | 0
  POL: 36 months, BL Yes (n=33,18) | 0 | 0
  POL: 36 months, BL No (n=33,18) | 1 | 0
  POL: 36 months, BL Missing (n=33,18) | 0 | 0
  FIB: 6 months post-treatment, BL Yes (n=16,17) | 1 | 0
  FIB: 6 months post-treatment, BL No (n=16,17) | 1 | 0
  FIB: 6 months post-treatment,BL Missing(n=16,17) | 0 | 2
  POL: 6 months post-treatment, BL Yes (n=16,17) | 0 | 0
  POL: 6 months post-treatment, BL No (n=16,17) | 0 | 0
  POL: 6 months post-treatment,BL Missing(n=16,17) | 1 | 0
  FIB: 12 months post-treatment, BL Yes (n=51,38) | 1 | 1
  FIB: 12 months post-treatment, BL No (n=51,38) | 2 | 0
  FIB: 12 months post-treatment, BL Missing(n=51,38) | 1 | 1
  POL: 12 months post-treatment, BL Yes (n=51,38) | 0 | 0
  POL: 12 months post-treatment, BL No (n=51,38) | 0 | 0
  POL: 12 months post-treatment, BL Missing (n=51,38 | 0 | 2
  FIB: 24 months post-treatment, BL Yes (n=43,31) | 2 | 2
  FIB: 24 months post-treatment, BL No (n=43,31) | 2 | 1
  FIB: 24 months post-treatment, BL Missing(n=43,31) | 1 | 2
  POL: 24 months post-treatment, BL Yes (n=43,31) | 0 | 0
  POL: 24 months post-treatment, BL No (n=43,31) | 1 | 0
  POL: 24 months post-treatment, BL Missing(n=43,31) | 2 | 1

27. Secondary Outcome: Percentage of Participants With at Least 1 Gynecological Symptoms: Endometrial Sub-study
Description: Gynecological symptoms included bleeding/spotting, pelvic pain, leucorrhoea and vaginal itching.
Time Frame: Baseline up to 24 months post-treatment
Population: As treated population included all treated participants, irrespective of the treatment duration and allocated to the group that corresponded to the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 86 | 94
percentage of participants | 16.28 | 21.28

28. Secondary Outcome: Number of Participants With Histological Findings: Endometrial Sub-study
Time Frame: Baseline up to 24 months post-treatment
Population: Results were not reported for this outcome measure because no data was collected as per change in planned analysis.
Arm/Group | Exemestane | Tamoxifen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: SAEs, AEs collected in separate databases.For SAE:treated population included all randomized participants with at least 1 study drug administration as per actual treatment received.For AE:safety population included all participants in treated population with at least 1 on-treatment AE assessment.AEs included AEs and illnesses reported during study.
Arm/Group | Exemestane | Tamoxifen
Serious Adverse Events (participants affected / at risk) | 383/2320 | 439/2338
Other Adverse Events (participants affected / at risk) | 1905/2249 | 1888/2279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=2320) | Tamoxifen (N=2338)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5
Acute myocardial infarction (Cardiac disorders) | 5 | 0
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 4 | 4
Angina unstable (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 8
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 6 | 2
Cardiac failure congestive (Cardiac disorders) | 5 | 3
Cardiac valve disease (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 2
Cyanosis (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 9 | 5
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Porphyria non-acute (Congenital, familial and genetic disorders) | 0 | 1
Auricular perichondritis (Ear and labyrinth disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Endocrine disorder (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 4 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 2
Eyelid ptosis (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1
Retinal vein thrombosis (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Diverticulitis oesophageal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 5
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 4 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 1 | 1
Axillary pain (General disorders) | 1 | 0
Chest pain (General disorders) | 5 | 4
Condition aggravated (General disorders) | 17 | 14
Death (General disorders) | 3 | 1
Device failure (General disorders) | 0 | 1
Disease progression (General disorders) | 4 | 10
Disease recurrence (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Gait disturbance (General disorders) | 0 | 1
Granuloma (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 1
Hyperplasia (General disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pelvic mass (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 4
Sudden death (General disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 3
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 7 | 9
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 2
Abdominal hernia gangrenous (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 3
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 5
Cellulitis laryngeal (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 3 | 1
Ear infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 4
Gastroenteritis (Infections and infestations) | 0 | 4
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 2
Mastitis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 4
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 4
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 4
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 3
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 7 | 8
Head injury (Injury, poisoning and procedural complications) | 0 | 3
Hip fracture (Injury, poisoning and procedural complications) | 4 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 3
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 4
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Retinal injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Calcification metastatic (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetic complication (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid intake reduced (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 14
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 17
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Axonal neuropathy (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 3
Carpal tunnel syndrome (Nervous system disorders) | 9 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 3 | 3
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 10 | 12
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 2
Encephalitis (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Hyperkinesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 3 | 3
Transient ischaemic attack (Nervous system disorders) | 4 | 7
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Catatonia (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 3 | 3
Hypomania (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 3
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 2
Colpocele (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 5
Ectropion of cervix (Reproductive system and breast disorders) | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 8
Endometrial hypertrophy (Reproductive system and breast disorders) | 2 | 5
Genital discharge (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 4 | 4
Ovarian cyst (Reproductive system and breast disorders) | 1 | 3
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 3
Rectocele (Reproductive system and breast disorders) | 1 | 3
Uterine disorder (Reproductive system and breast disorders) | 0 | 2
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 3 | 25
Uterine prolapse (Reproductive system and breast disorders) | 3 | 6
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 7 | 11
Vaginal prolapse (Reproductive system and breast disorders) | 2 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Bone graft (Surgical and medical procedures) | 0 | 1
Breast lump removal (Surgical and medical procedures) | 1 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 1 | 2
Breast prosthesis removal (Surgical and medical procedures) | 0 | 1
Breast reconstruction (Surgical and medical procedures) | 2 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 3 | 1
Dacryocystorhinostomy (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 2 | 5
Hysterectomy (Surgical and medical procedures) | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 3
Knee operation (Surgical and medical procedures) | 1 | 0
Laparotomy (Surgical and medical procedures) | 0 | 1
Maxillofacial operation (Surgical and medical procedures) | 0 | 1
Meniscus operation (Surgical and medical procedures) | 0 | 1
Nasal septal operation (Surgical and medical procedures) | 0 | 1
Plastic surgery (Surgical and medical procedures) | 1 | 0
Prosthesis implantation (Surgical and medical procedures) | 1 | 0
Scar excision (Surgical and medical procedures) | 0 | 2
Skin graft (Surgical and medical procedures) | 1 | 1
Surgery (Surgical and medical procedures) | 3 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 2
Vaginoplasty (Surgical and medical procedures) | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 0 | 1
Vitrectomy (Surgical and medical procedures) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 4 | 22
Haematoma (Vascular disorders) | 2 | 1
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 8 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 2
Phlebitis superficial (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 3
Thrombophlebitis superficial (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=2249) | Tamoxifen (N=2279)
Nausea (Gastrointestinal disorders) | 200 | 208
Fatigue (General disorders) | 367 | 344
Weight increased (Investigations) | 128 | 138
Arthralgia (Musculoskeletal and connective tissue disorders) | 396 | 246
Back pain (Musculoskeletal and connective tissue disorders) | 208 | 176
Osteoarthritis NOS (Musculoskeletal and connective tissue disorders) | 138 | 106
Osteoporosis NOS (Musculoskeletal and connective tissue disorders) | 116 | 66
Pain in limb (Musculoskeletal and connective tissue disorders) | 143 | 108
Dizziness (Nervous system disorders) | 224 | 200
Headache (Nervous system disorders) | 305 | 255
Depression (Psychiatric disorders) | 140 | 127
Insomnia (Psychiatric disorders) | 290 | 205
Vaginal haemorrhage (Reproductive system and breast disorders) | 89 | 121
Sweating increased (Skin and subcutaneous tissue disorders) | 270 | 242
Hot flushes NOS (Vascular disorders) | 491 | 457
Hypertension NOS (Vascular disorders) | 223 | 191

LIMITATIONS AND CAVEATS:
Other AEs included both SAEs and AEs. Non-SAE could not be presented separately for this study as AEs were collected in clinical database where SAE flags were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.